CLINICAL TRIAL: NCT05536635
Title: The Effect of Breathing Techniques on Attack Frequency and Severity in Migraine-like Headaches-randomised Control Trial: Study Protocol for a Cluster Randomised Controlled Trial
Brief Title: Effect of Breathing Techniques on Migraine Attacks and Severity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Oğulcan Çöme, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7201
Record Dates: First submitted 2022-09-06; First posted 2022-09-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Migraine Headaches; Breathing Techniques
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- breathing techniques (Experimental): The patients in the intervention group will be taught and practiced breathing technique. Breathing techniques will be taught face-to-face by the researcher to the patients in the intervention group. The participant will breathe through one nostril at a natural rate and depth, while the other nostril will be closed with the thumb or forefinger. After the act of breathing, it will open the closed nostril, close the open nostril and breathe naturally. As explained later, they will continue the cycle with the act of breathing. This process is described as a loop.
  Interventions: Behavioral: breathing techniques
- treatment as usual (No Intervention): The control group will continue his/her usual treatment as advised by the physician.

INTERVENTIONS:
Behavioral: breathing techniques — Intervention will be daily use of breathing techniques thought by the researcher as explained in detail in arm/group descriptions
  Arms: breathing techniques

SUMMARY:
Background:

Migraine is a very common neurobiological disorder caused by increased excitability of the Central Nervous System. It is among the causes of the highest morbidity worldwide. Migraine has considerable economic and social impact ; affects the quality of life of patients and disrupts work life, social activities and family life. To decrease the frequency and severity of migraine attacks may be the first goal than treating the attacks.

The study was designed as a Parallel Group, Add on, Randomized Controlled Experiment in order to observe the effects of breathing techniques on migraine-like headaches, frequency and severity.

Methods:

Participants will be divided into 2 parallel arms, intervention and control (treatment as usual). Cluster randomization will be performed to prevent intergroup contamination. Breathing techniques will be taught to the intervention group by the researcher. Both groups will continue to use pharmacotherapy for migraine. Both groups will be evaluated with migraine disability level (MIDAS) at the beginning and end of the study. The primary output of the study is to evaluate the effect of breathing techniques on the frequency and severity of attacks in migraine-like headaches. The secondary output is to evaluate the effect of breathing techniques on the MIDAS level.

Discussion:

The results of the study will provide information about the effect of breathing techniques on migraine-like headaches. The results of this study will contribute to the literature, since migraine is among the chronic diseases and pharmacotherapy options are limited.

ELIGIBILITY:
Inclusion Criteria:

* Are 18-50 Age
* Have a computer and/or smart phone
* Have an internet connection that can be used at home and at work (with a computer or smart phone)
* Are volunteer to participate in the research
* Have Frequency of attacks less than 3 months
* Fulfil diagnostic criteria of migraine like headaches

Exclusion Criteria:

* Severe anatomical defect in the airway
* Pregnancy
* Having any diagnosed psychiatric disease
* Using psychiatric medication
* Having speech and hearing problems
* Having any chronic disease which may be worsening by taking deep breath

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Determining effects of breathing techniques on migraine like headaches frequency and intensity with "migraine disability assessment " (MIDAS) questionnaire. | Three months
  The MIDAS is a self-administered tool to assess migraine-related disability over the previous 3 months . The questionnaire comprises seven questions in total. Three questions assess the number of missed days due to headache. Two questions assess the number of additional days with limited productivity. The total MIDAS score is the sum of the days given as response to these five questions. The total score ranges from 0 to 90 and is used to categorize patients in disability grades I to IV. A higher score means more severe disability.Two additional questions measure headache frequency and average pain intensity. Frequency is noted as the number of days in the previous 3 months on which the patient experienced migraine. Intensity is noted as the average pain intensity of these episodes on a scale of 1-10. These two items are not taken into account when estimating the total MIDAS score.

SECONDARY OUTCOMES:
Determining effects of breathing techniques to "migraine disability assessment " (MIDAS) scores of migraine patients. | Three months
  The MIDAS is a self-administered tool to assess migraine-related disability over the previous 3 months . The questionnaire comprises seven questions in total. Three questions assess the number of missed days due to headache. Two questions assess the number of additional days with limited productivity. The total MIDAS score is the sum of the days given as response to these five questions. The total score ranges from 0 to 90 and is used to categorize patients in disability grades I to IV. A higher score means more severe disability.Two additional questions measure headache frequency and average pain intensity. Frequency is noted as the number of days in the previous 3 months on which the patient experienced migraine. Intensity is noted as the average pain intensity of these episodes on a scale of 1-10. These two items are not taken into account when estimating the total MIDAS score.

CONTACTS AND LOCATIONS:
Overall Officials: ogulcan D come, MD, Principal Investigator — Dokuz Eylul University Medical School
Locations (1):
- Dokuz Eylul University Faculty of Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silberstein SD. Migraine. Lancet. 2004 Jan 31;363(9406):381-91. doi: 10.1016/S0140-6736(04)15440-8. PMID 15070571
- [Background] Burch R, Rizzoli P, Loder E. The Prevalence and Impact of Migraine and Severe Headache in the United States: Figures and Trends From Government Health Studies. Headache. 2018 Apr;58(4):496-505. doi: 10.1111/head.13281. Epub 2018 Mar 12. PMID 29527677
- [Background] Ciarambino T, Sansone G, Menna G, Para O, Signoriello G, Leoncini L, Giordano M. Oxygen Therapy in Headache Disorders: A Systematic Review. Brain Sci. 2021 Mar 17;11(3):379. doi: 10.3390/brainsci11030379. PMID 33802647
- [Background] Bennett MH, French C, Schnabel A, Wasiak J, Kranke P. Normobaric and hyperbaric oxygen therapy for migraine and cluster headache. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD005219. doi: 10.1002/14651858.CD005219.pub2. PMID 18646121
- [Background] Singhal AB, Maas MB, Goldstein JN, Mills BB, Chen DW, Ayata C, Kacmarek RM, Topcuoglu MA. High-flow oxygen therapy for treatment of acute migraine: A randomized crossover trial. Cephalalgia. 2017 Jul;37(8):730-736. doi: 10.1177/0333102416651453. Epub 2016 May 20. PMID 27206964
- [Background] Matera DV, Smith B, Lam B. Revisiting the expanded use of hyperbaric oxygen therapy for treatment of resistant migraines. Med Gas Res. 2019 Oct-Dec;9(4):238-240. doi: 10.4103/2045-9912.273963. PMID 31898611
- [Background] Bernardi L, Spadacini G, Bellwon J, Hajric R, Roskamm H, Frey AW. Effect of breathing rate on oxygen saturation and exercise performance in chronic heart failure. Lancet. 1998 May 2;351(9112):1308-11. doi: 10.1016/S0140-6736(97)10341-5. PMID 9643792
- [Background] Bilo G, Revera M, Bussotti M, Bonacina D, Styczkiewicz K, Caldara G, Giglio A, Faini A, Giuliano A, Lombardi C, Kawecka-Jaszcz K, Mancia G, Agostoni P, Parati G. Effects of slow deep breathing at high altitude on oxygen saturation, pulmonary and systemic hemodynamics. PLoS One. 2012;7(11):e49074. doi: 10.1371/journal.pone.0049074. Epub 2012 Nov 12. PMID 23152851
- [Background] Russo MA, Santarelli DM, O'Rourke D. The physiological effects of slow breathing in the healthy human. Breathe (Sheff). 2017 Dec;13(4):298-309. doi: 10.1183/20734735.009817. PMID 29209423
- [Background] Spatenkova V, Bednar R, Oravcova G, Melichova A, Kuriscak E. Yogic breathing in hypobaric environment: breathing exercising and its effect on hypobaric hypoxemia and heart rate at 3,650-m elevation. J Exerc Rehabil. 2021 Aug 23;17(4):270-278. doi: 10.12965/jer.2142324.162. eCollection 2021 Aug. PMID 34527639
- [Background] Moher D, Jones A, Lepage L; CONSORT Group (Consolidated Standards for Reporting of Trials). Use of the CONSORT statement and quality of reports of randomized trials: a comparative before-and-after evaluation. JAMA. 2001 Apr 18;285(15):1992-5. doi: 10.1001/jama.285.15.1992. PMID 11308436
- [Background] Campbell MK, Elbourne DR, Altman DG; CONSORT group. CONSORT statement: extension to cluster randomised trials. BMJ. 2004 Mar 20;328(7441):702-8. doi: 10.1136/bmj.328.7441.702. No abstract available. PMID 15031246
- [Background] Campbell MJ, Donner A, Klar N. Developments in cluster randomized trials and Statistics in Medicine. Stat Med. 2007 Jan 15;26(1):2-19. doi: 10.1002/sim.2731. PMID 17136746
- [Background] Roberts C, Roberts SA. Design and analysis of clinical trials with clustering effects due to treatment. Clin Trials. 2005;2(2):152-62. doi: 10.1191/1740774505cn076oa. PMID 16279137